CLINICAL TRIAL: NCT07265986
Title: Comparison Between a Robotic Tele-echo-cardiography Technique and a Standard Echocardiography in the Management of Heart Failure in the Guadeloupe Archipelago Between the University Hospital of Guadeloupe and the Marie-Galante Hospital
Acronym: TER de blueS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Collaborators: GIRCI SOHO (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: PAP_RI2_2019/02
Record Dates: First submitted 2025-11-14; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure; Remote Consultation, Teleconsultation; Echocardiography, Doppler
Keywords: heart failure; remote echocardiography doppler; telemedicine
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: This is a prospective multicentre study (one cardiologist in a private practice in Guadeloupe and one at the Marie-Galante Hospital) interventional cross-over study in which the measurements obtained successively by tele-echo-cardiography and standard echocardiography will be compared. Among the set of parameters to be measured, we have chosen the left ventricular ejection fraction (LVEF) as the main judgement criterion because this measure defines the type of heart failure.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: in situ ultrasound (EIS) performed first (Experimental): The in situ ultrasound (EIS) is performed first. Cardiologist A performs the imaging examination and then leaves the room. The Research Nurse installs the probe and then cardiologist B, positioned on the expert site in Guadeloupe, carries out the examination of robotic tele-echo-cardiography (TER). Cardiologist B communicates via videoconferencing with the patient and the Research Nurse.
  Interventions: Diagnostic Test: in situ echocardiography (EIS); Diagnostic Test: two-dimensional remote echocardiography (TER)
- Arm B: two-dimensional remote echocardiography (TER) performed first (Experimental): The TER is carried out first. The probe is installed by the REsearch Nurse, cardiologist B positioned on the expert site of Guadeloupê carries out the TER examination. Cardiologist B communicates via videoconferencing with the patient and the remote assistant EDI. Then, once the examination is completed, cardiologist A performs the HIA.
  Interventions: Diagnostic Test: in situ echocardiography (EIS); Diagnostic Test: two-dimensional remote echocardiography (TER)

INTERVENTIONS:
Diagnostic Test: in situ echocardiography (EIS) — In situ echocardiography (EIS) will be performed by the cardiologist present in Marie-Galante Hospital.
Diagnostic Test: two-dimensional remote echocardiography (TER) — Remote echocardiography is performed by a cardiologist from a private practice in Guadeloupe, with a research nurse present at the patient's side at Marie-Galante Hospital.

SUMMARY:
The TERdeblue-S study is a feasibility study of robotic remote echocardiography, not only in terms of technology but also in terms of its integration into a telemedicine system to improve access to the heart failure management system in the Guadeloupe archipelago. The main objective of this study is to study the agreement of the measurement of the left ventricular ejection fraction (FejVG) between in situ echocardiography (EIS) and two-dimensional remote echocardiography (TER) (distance and volumes).

DETAILED DESCRIPTION:
Considered as the new global epidemic of the 21st century, heart failure (HF) is a major public health issue. In 2010, the Guadeloupe region already had the highest rate of heart failure deaths in all French departments, furthermore cardiac decompensation of chronic heart failure is the first cardiovascular pathology to be managed in emergency medicine and the first cardiovascular cause of hospitalization. Marie-Galante is an island in the Guadeloupe archipelago, 36% of whose hospital stays are covered by the University Hospital Currently, access to specialized care in Marie-Galante, particularly cardiological care, is very limited with one to two monthly consultations by a specialist cardiologist accessible to a population . Rather, remote echocardiography has been the subject of experimental studies but has not yet been proposed as part of an optimization of the management of a specific cardiovascular disease at separate sites. This is a prospective multicentre study (two cardiologists in private practice of Guadeloupe and one at the Marie-Galante Hospital) interventional cross-over study in which the left ventricular ejection fraction (LVEF) will be the main judgement criterion. Patients will be randomized to determine the order of implementation of the techniques (echocardiography and then teleecardiography or the reverse). In addition, in order to take into account the operator effect, each of the 2 cardiologists will move alternately either for remote echocardiography or to Marie-Galante for in situ echocardiography.

The visit (V1) takes place at Marie-Galante's CH, as soon as possible after inclusion by the generalist practicionner or the cardiologist (V0) and is carried out by the state-registered nurse with a blood sample (biological check-up and biological collection) and ECG Holter place over 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years

  * Free, informed and written consent signed by the participant and the investigator
  * Person affiliated or benefiting from a social security scheme.
  * Patient meeting at least one of the following criteria:
* Systematic cardiovascular check-up or asymptomatic patient with cardiovascular risk factor (hypertension, diabetes, obesity, tobacco, alcohol)
* Clinical suspicion of heart disease and/or chronic heart failure with stability of at least one week.

  * Family history of heart disease and/or sudden death

Exclusion Criteria:

* Patient requiring urgent cardiological management with transfer to the University Hospital

  * Acute unstable heart failure, admission to CH Marie-Galante less than 5 days (less than one week)
  * Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11-30 (Actual); Primary Completion 2026-09-08 (Estimated); Study Completion 2026-09-08 (Estimated)

PRIMARY OUTCOMES:
Agreement of Left Ventricular Ejection Fraction (LVEF) Measurements Between Echocardiography Techniques | Measured at the second visit (V2) at 2 weeks.
  The main outcome measure is the agreement of left ventricular ejection fraction (LVEF) measurements between two echocardiography techniques. Agreement will be quantified using the intraclass correlation coefficient (ICC) and supplemented by Bland-Altman plots to visualize differences between methods.

SECONDARY OUTCOMES:
Agreement Between Echocardiography Techniques for Diagnosis of Cardiac Anomalies | Measured at the second visit (V2) at 2 weeks.
  Agreement between two echocardiography techniques for diagnosing cardiac anomalies (dilated cardiomyopathy, hypertrophic cardiomyopathy, and valvulopathies) will be evaluated using the Kappa coefficient. Sensitivity and specificity of each technique for each anomaly will also be reported.
Dilated Cardiomyopathy Assessment | Measured at Visit 2 (V2), 2 weeks after baseline.
  Presence or absence of dilated cardiomyopathy will be defined according to left ventricular telediastolic diameter and reported as number of participants with dilated cardiomyopathy for each technique.
Quantitative Echocardiographic Measures | Measured at the second visit (V2) at 2 weeks.
  Agreement between the two echocardiography techniques will be assessed using the intraclass correlation coefficient (ICC), paired Student's t-test, and Bland-Altman plots for the following measures:
  Diastolic function - mitral Doppler inflow/outflow (I/O) ratio and tissue Doppler I/O ratio; Aortic flow - measured from subaortic velocity-time integral (ITV); Systolic pulmonary arterial pressure - derived from tricuspid insufficiency using the Bernoulli formula; Right ventricular systolic function - assessed by TAPSE.
Hypertrophic Cardiomyopathy Assessment | Measured at Visit 2 (V2), 2 weeks after baseline.
  Presence or absence of hypertrophic cardiomyopathy will be defined based on septal and posterior wall thickness and reported as number of participants with hypertrophic cardiomyopathy for each technique.
Valvulopathy Assessment | Measured at V2 (2 weeks)
  Presence or absence of aortic or mitral stenosis and regurgitation will be reported as number of participants with valvulopathies for each technique.
Systolic Pulmonary Arterial Pressure (PAP) | Measured at V2 (2 weeks)
  Systolic PAP will be measured from tricuspid regurgitation or estimated indirectly from systolic pulmonary ejection flow. Reported in mmHg.
Left Ventricular Filling Pressure | Measured at V2 (2 weeks)
  Changes in left ventricular (LV) filling pressures will be assessed using the E/e' ratio (mitral Doppler flow / tissue Doppler flow at the mitral annulus).
Duration of Echocardiography | Measured at the second visit (V2) at 2 weeks.
  Total duration of each echocardiography session will be recorded in minutes for both techniques.
Patient Satisfaction | Measured at the second visit (V2) at 2 weeks.
  Patient satisfaction with the tele-echocardiography procedure will be assessed using an adapted TeleHealth Satisfaction Questionnaire (TSQ).
  Each item is scored on a 5-point Likert scale (1 = very dissatisfied, 5 = very satisfied), resulting in a total score range of 0 to 100 after standardization, where higher scores indicate greater satisfaction.
  All assessments will be conducted at the tele-echocardiography session by a blinded evaluator or self-reported by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Mona Hedreville, MD, Study Chair
Locations (3):
- Guadeloupe (3):
  - Centre Hospitalier Sainte-Marie de Marie-Galante, Grand-Bourg
  - Centre de Cardiologie Zac Colin, Petit-Bourg
  - Cabinet de cardiologie TONCOEURTONKA, Petit-Canal

IPD SHARING:
Plan to Share IPD: No